CLINICAL TRIAL: NCT00003394
Title: Phase I/II Study of Weekly Intravenous Estramustine Phosphate in Combination With Paclitaxel and Carboplatin in Patients With Advanced Prostate Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-032; CDR0000066392 (Registry Identifier: PDQ (Physician Data Query)); NCI-G98-1448
Record Dates: First submitted 1999-11-01; First posted 2004-04-30 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Carboplatin; Estramustine; Goserelin; Leuprolide; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: endocrine-modulating drug therapy
Drug: estramustine phosphate sodium
Drug: goserelin acetate
Drug: leuprolide acetate
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy consisting of estramustine, paclitaxel, and carboplatin in treating patients with advanced prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine a safe weekly dose of intravenous estramustine (EM) in combination with paclitaxel (TAX) and carboplatin (CBDCA) in patients with advanced prostate cancer. II. Determine the safety and efficacy of this combination in androgen dependent vs androgen independent disease in these patients. III. Evaluate the pharmacokinetics of weekly intravenous EM and TAX in combination with CBDCA in these patients.

OUTLINE: Phase I is a dose escalation study of estramustine. Phase II is a two stage design study, in which patients are stratified according to androgen dependence (androgen dependent disease vs androgen independent disease). In phase I, patients receive estramustine IV over 1 hour via permanent venous access device on day 1 of weeks 1, 2, 3, and 4, followed by paclitaxel (TAX) IV over 1 hour. Carboplatin IV is administered over 30 minutes at the completion of TAX at week 1. Courses repeat every 4 weeks until disease progression or excessive toxicity or for up to 24 weeks. Patients with locally advanced androgen dependent prostate cancer may be considered for radical prostatectomy or radiotherapy after 4 courses. Androgen dependent patients not already on primary hormone therapy with a GnRH analog receive goserelin or leuprolide injections under the skin every 3 months while on the study, beginning during the first or second week of therapy. Three patients are entered at each dose level and must complete one course of therapy. If no patient experiences dose limiting toxicity (DLT), then 3 patients are treated at the next higher dose level. If 1 patient experiences DLT, then 3 more patients are treated at that same dose level. If 2 of 6 patients experience DLT, then that dose is declared the maximum tolerated dose (MTD). In phase II, a two stage design is applied to each patient population. Fourteen patients are enrolled in the first stage. If no responses are observed, the trial is stopped. If at least 1 response is observed, 11 additional patients will be enrolled onto the study.

PROJECTED ACCRUAL: A total of 6-18 patients will be accrued to phase I; phase II will accrue up to 50 patients within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven prostate cancer that is androgen dependent or independent Androgen dependent disease must meet ONE OR MORE of the following criteria: (1) Previously untreated, locally advanced adenocarcinoma of the prostate and: T1-2 tumor stage, PSA greater than 20 ng/mL OR T3-4 tumor stage OR Gleason grade 8-10 (2) Small cell carcinoma, poorly differentiated tumor with neuroendocrine features, or neuroendocrine carcinoma of any stage (3) Disease metastatic to bones or soft tissues (visceral or lymph nodes) that is evaluable on MRI, CT, or bone scan (patients with evaluable disease that relapsed after neoadjuvant hormone therapy prior to radical prostatectomy or radiotherapy are eligible) Patients meeting one of the above criteria who have started on an antiandrogen (flutamide, nilutamide, or bicalutamide) and/or a gonadotropin releasing hormone (GnRH) analog (luprolide or goserelin) are eligible if they have been on androgen ablation (GnRH analog with or without antiandrogen) for no more than 3 months Androgen independent disease must meet ALL of the following criteria: (1) Disease progression despite primary hormone treatment (e.g., orchiectomy, estrogen therapy, GnRH analog with or without an antiandrogen), OR disease progression despite receiving antiandrogen treatment as part of primary hormone therapy, evidenced by: Bone (new osseous lesion) or Soft tissue (greater than 25% increase in bidimensionally measurable disease) or Rising PSA (on any 3 determinations taken at weekly intervals (at least) to greater than 50% above the patient's baseline PSA value) despite castrate (no greater than 30 ng/mL) levels of testosterone (2) At least 2 weeks since change in hormone therapy (including prednisone or dexamethasone) (3) Continuation on treatments to maintain castrate levels of testosterone if no prior orchiectomy (4) Evaluable or measurable disease (5) No more than 1 prior course of chemotherapy (6) No more than 1 prior course of palliative radiotherapy or radioisotope treatment (strontium chloride Sr 89)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 120,000/mm3 Hemoglobin at least 8.0 g/dL Hepatic: Bilirubin no greater than 1.5 mg/dL or 1.5 times upper limit of normal (ULN) AST no greater than 56 U/L or 1.5 times ULN Renal: Creatinine no greater than 2.0 mg/dL or 1.5 times ULN Cardiovascular: At least 6 months since acute deep vein thrombosis and/or pulmonary embolism No serious ventricular arrhythmia No significant heart disease No active angina (stable or unstable) No myocardial infarction within 6 months No congestive heart failure No transient ischemic attack or stroke within 6 months Neurologic: No grade 3-4 peripheral neuropathy Other: No severe infection No severe malnutrition No other serious medical illnesses

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since immunotherapy Chemotherapy: See Disease Characteristics At least 4 weeks since chemotherapy No other concurrent chemotherapy Endocrine therapy: See Disease Characteristics Radiotherapy: See Disease Characteristics At least 4 weeks since radiotherapy (8 weeks if systemic radioisotope treatment with strontium chloride Sr 89) No concurrent radiation of the only measurable lesion No concurrent radiotherapy or radioisotope therapy Surgery: See Disease Characteristics At least 4 weeks since major surgery No concurrent surgery to the only measurable lesion Other: Permanent venous access device (e.g., mediport or Hickman catheter) required

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 1998-04; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William K. Kelly, DO, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States